CLINICAL TRIAL: NCT05884073
Title: The Cost of Caring: Examining the Role of Exercise in Mitigating Oncology Care Provider Burnout (C4C+)
Brief Title: Exercise for Oncology Care Professionals
Acronym: C4C+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melanie Keats (Other)
Responsible Party: Sponsor-Investigator, Melanie Keats, Principal Investigator, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C4C+
Record Dates: First submitted 2023-05-05; First posted 2023-06-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Burnout, Caregiver; Compassion Fatigue
Keywords: oncology health professionals; burnout; exercise; physical activity; nature-based walking
MeSH Terms: conditions — Caregiver Burden; Compassion Fatigue; Burnout, Psychological; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circuit-based resistance exercise (Experimental): 12-week, supervised circuit-based resistance training program (2-3 times/week).
  Interventions: Behavioral: Circuit-based Resistance Training
- Nature Walking (Active Comparator): 12-weeks self-paced walking in nature (2-3 times/week).
  Interventions: Behavioral: Nature-based Walking

INTERVENTIONS:
Behavioral: Circuit-based Resistance Training — Participants will engage in a 12-week circuit-based resistance training program 2-3 times/week. Each supervised session will last about 30 minutes and will consist of 5 resistance exercises. Each exercise will be completed for 1 minute for a total of 5 minutes followed by a 1-minute rest. The circuit will then repeated 3 additional times (total of 4 circuits). All resistance sessions will be supervised by a certified fitness professionals.
  Arms: Circuit-based resistance exercise
Behavioral: Nature-based Walking — Participants will be asked to engage in 30 minutes of self-paced walking in nature 2-3 days/week. Participants will be provided with a list of resources that direct them to walkable nature/green spaces close to their home or workplace.
  Arms: Nature Walking

SUMMARY:
The goal of this preference-based pilot study will be to assess the feasibility and acceptability, and impact of a 12-week exercise intervention on oncology care provider burnout. Participants self-select to participate into one of two exercise groups. Group assignment will be based on participant preference.

Group 1: Supervised circuit-based resistance exercise

Group 2: Nature-based walking

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Able to speak/write in English;
* Must be providing formal care to cancer patients in a clinical setting within the Halifax Municipality;
* Actively practicing within the Nova Scotia Cancer Care Program; and
* Able and willing to engage in low-to-moderate intensity physical activity.

Exclusion Criteria:

* Exceeding Canadian physical activity guidelines of 150-minutes of moderate-to-vigorous physical activity per week; and
* Any health condition that would preclude safe participation in a new exercise program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Participant Fidelity (Intervention Adherence) | Through study completion (about 2 years)
  Participant adherence to prescribed exercise intervention
Feasibility - Safety | Through study completion (about 2 years)
  Adverse and serious adverse events
Feasibility - Retention/Attrition | Through study completion (about 2 years)
  Percentage of participants who complete the 12-week intervention
Feasibility - Attendance | Through study completion (about 2 years)
  Attendance is calculated as the percentage of exercise sessions completed by the total number of available exercise sessions over the 12-week intervention.
Feasibility - Recruitment | Through study completion (about 2 years)
  Participant accrual as defined as the number of eligible participants who express an interest in participation divided by the number of participants who consent to participate.
Feasibility - Participant Experience | Through study completion (about 2 years)
  Interviews with a diverse group of participants will be used to assess factors influencing participant selection of intervention type/setting, adherence to and satisfaction with the selected intervention.

SECONDARY OUTCOMES:
Maslach Burnout Inventory (MBI) for Medical Personnel (MP) | Baseline, mid-program (6-weeks), and post intervention (12-weeks).
  The MBI-MP is used to assess burnout in medical professionals. The 22-item, 7-point Likert scale (0 = never to 6 = everyday) assesses burnout across three dimensions: emotional exhaustion (9 items), personal accomplishment (8 items), and depersonalization (5-items).
Physical Activity Behavior - Self-reported | Baseline, mid-program (6-weeks), and post intervention (12-weeks).
  Self-reported physical activity is assessed by the Godin Leisure Time Exercise Questionnaire. Higher scores indicate higher levels of physical activity. Participants reporting moderate-to-strenuous Leisure Score Index ≥ 24 are classified as active; those reporting moderate-to-strenuous Leisure Score Index ≤ 23 are classified as insufficiently active.
Resting heart rate | Pre to post intervention (12-week change)
  Resting heart rate
Resting Blood Pressure | Pre to post intervention (12-week change)
  Resting systolic and diastolic blood pressure
Aerobic fitness | Pre to post intervention (12-week change)
  The six-minute walk test is used to assess aerobic capacity.
Upper Body Strength | Pre to post intervention (12-week change)
  A hand-held dynamometer is used to assess upper body strength.
Muscular Endurance | Pre to post intervention (12-week change)
  The 30-second sit-to-stand is used to assess lower body muscular endurance.
Body Mass Index | Pre to post intervention (12-week change)
  Height and weight is used to assess body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Activity and Cancer (PAC) Lab, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No